CLINICAL TRIAL: NCT04473417
Title: An Open-label, Randomized, Single-dose, Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of DA-2811 in Healthy Subjects
Brief Title: Pharmacokinetics and Safety/Tolerability Profiles of DA-2811 in Healthy Subjects
Acronym: DA-2811
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA2811_BE_I
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A, Sequence I (Experimental): Period I: Forxiga® → DA-2811, Period II: DA-2811 → Forxiga®
  Interventions: Drug: Forxiga; Drug: DA-2811
- Part A, Sequence II (Experimental): Period I: DA-2811 → Forxiga®, Period II: Forxiga® → DA-2811
  Interventions: Drug: Forxiga; Drug: DA-2811
- Part B, Sequence I (Experimental): Period I: DA-2811 under fasting state → DA-2811 under fed state, Period II:DA-2811 under fed state → DA-2811 under fasting state
  Interventions: Drug: DA-2811
- Part B, Sequence II (Experimental): Period I: DA-2811 under fed state → DA-2811 under fasting state, Period II: DA-2811 under fasting state → DA-2811 under fed state
  Interventions: Drug: DA-2811

INTERVENTIONS:
Drug: Forxiga — single dose administration after 10hr fasting
  Arms: Part A, Sequence I; Part A, Sequence II
Drug: DA-2811 — single dose administration after 10hr fasting
  Arms: Part A, Sequence I; Part A, Sequence II
Drug: DA-2811 — single dose administration after 10hr fasting
  Arms: Part B, Sequence I; Part B, Sequence II
Drug: DA-2811 — single dose administration after high fat and calorie fed diet
  Arms: Part B, Sequence I; Part B, Sequence II

SUMMARY:
This is the phase I study to evaluate the pharmacokinetics and safety of DA-2811 and Forxiga® after a single oral dose in healthy volunteers.

The study will also compare the pharmacokinetics and safety profiles of DA-2811 under fasting and fed states in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects
* BMI between 18.5 and 29.9 kg/m2 and weigh at least 50 kg
* Volunteer who totally understands the progress of this clinical trial, make decision by his or her free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Volunteer who has present or past history of clinically significant cardiovascular, respiratory, urinary, gastrointestinal, hepatic, renal, skin, immunological, musculoskeletal, endocrinal, neurological, psychiatric and/or hematological disease
* Vulnerable to dehydration due to poor oral intake or clinically significant dehydration as judged by the investigator
* History of gastrointestinal disease or any gastrointestinal surgery(except for simple appendectomy, hernia surgery, hemorrhoid surgery)
* History of diseases that may impact absorption, distribution, metabolism, and excretion of the study drugs.
* Hypersensitivity to a drug containing an ingredient of the investigational product, Sodium glucose transporter-2 inhibitors, additional ingredient or other drugs (e.g., aspirin, antibiotics, etc.) or medical history of clinically significant hypersensitivity.
* History of clinically significant active chronic disease
* volunteer who has genetic disorder like lapp lactase deficiency or glucose-galactose malabsorption.
* History of clinically significant allergies including drug allergies
* History of drug abuse or addicted
* Clinical laboratory test values are outside the accepted normal range
* Participation in another clinical trial within 6 months of the first IP administration
* Sexually active women of childbearing potential not consistently and correctly practicing birth control by dual contraceptive method until 2 months after last IP administration
* Breast-feeding period, pregnant, or positive to urine pregnancy test (conducted before the first drug administration)
* Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
AUClast | pre-dose~48 hours post-dose
  Area under the plasma concentration-time curve from time zero to time the last quantifiable time
Cmax | pre-dose~48 hours post-dose
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUC(0 - ∞) | pre-dose~48 hours post-dose
  Area under the plasma concentration versus time curve from time zero to extrapolated infinite time (0 - ∞)
Tmax | pre-dose~48 hours post-dose
  Time to reach maximum plasma concentration following drug administration
t1/2 | pre-dose~48 hours post dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: JaeYong Chung, Principal Investigator — Bundang Seoul National University Hospital Clinical Trial Center
Locations (1):
- Bundangseoul national unversity hospital, Sŏngnam, GyeonggiDo, South Korea